CLINICAL TRIAL: NCT01185678
Title: Observation of Compliance With Dosage in Women Using Oral Contraceptives Designed for the Non Stop Use, (it Means 28 Pills for 28-days Cycle).
Brief Title: Data on Oral Contraceptives Compliance in Non Stop Regimen
Acronym: DOC Non Stop
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Medical Director, Bayer Sp. z o.o.
Other Study IDs: 15253; WH1011PL (Other: Company internal)
Record Dates: First submitted 2010-08-19; First posted 2010-08-20 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2013-06

CONDITIONS: Contraception
Keywords: Contraception; Compliance
MeSH Terms: conditions — Patient Compliance | interventions — drospirenone and ethinyl estradiol combination; Contraceptives, Oral, Combined; Desogestrel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group1
  Interventions: Drug: Qlaira or Yaz (BSP products defined as Combined Oral Contraceptive) and Cerazette or Azalia (competitor's products defined as Progestogen Only Pill)

INTERVENTIONS:
Drug: Qlaira or Yaz (BSP products defined as Combined Oral Contraceptive) and Cerazette or Azalia (competitor's products defined as Progestogen Only Pill) — One tablet per day, orally, 28 tablets per cycle, during three consecutive cycles.

SUMMARY:
Adherence to the dosing scheme is the principal element of COC efficiency. On the other hand noncompliance seemed to be an inseparable element of any oral treatment. The aim of the study is to evaluate in everyday practice the relation between dosage errors and indicated factors, potentially influencing the compliance with the dosing scheme.

ELIGIBILITY:
Inclusion Criteria:

* Patients at the age of 18-50 requiring contraception, treated with oral contraceptives designed for the scheme 28 pills for 28 days. The decisions would be made at the discretion of the attending physician.

Exclusion Criteria:

* Patients were not valid for analysis if the initial visit was before start of study in the country (retrospective documentation), or if they did not take oral contraceptives designed for the scheme 28 pills for 28 days.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Gynecological practices ptients - starters or current users.
Sampling Method: Probability Sample
Enrollment: 8416 (Actual)
Dates: Start 2010-05; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
The percentage of users showing noncompliant behaviors | 3 consecutive cycles (28-days per cycle)

SECONDARY OUTCOMES:
The characteristics of noncompliant behavior. | 3 consecutive cycles (28-days per cycle)
The relation between noncompliant behavior and selected factors. | 3 consecutive cycles (28-days per cycle)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Poland